CLINICAL TRIAL: NCT03876301
Title: A Multi-Center, Observational Study in Males With Hemophilia A
Brief Title: Lead-in Study to Collect Prospective Efficacy and Safety Data of Current FVIII Prophylaxis Replacement Therapy in Adult Hemophilia A Participants
Status: Completed | Type: Observational
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPK-8011-301
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Blood Coagulation Disorder; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemophilia A; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Hematologic Diseases; Hemorrhagic Disorders; Factor VIII Deficiency
Keywords: Factor VIII; Factor VIII Protein; Recombinant
MeSH Terms: conditions — Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemophilia A; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Hematologic Diseases; Hemorrhagic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: Adult males with clinically severe hemophilia A, who are negative for neutralizing antibody (NAb) to AAV-Spark200
  Interventions: Drug: Standard of Care FVIII Replacement therapy

INTERVENTIONS:
Drug: Standard of Care FVIII Replacement therapy — There is no investigational product being administered. Subjects will be administering their own standard of care FVIII replacement therapy.

SUMMARY:
The aim of this prospective, observational study is to establish a dataset on the frequency of bleeding events, as well as other characteristics of bleeding events and FVIII infusions, in patients with clinically severe hemophilia A receiving prophylactic FVIII replacement therapy as standard of care. The data collected from this study may assist in providing baseline information for comparison to the Spark's investigational hemophilia A gene therapy in future Phase 3 studies.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Males ≥18 years of age.
3. Clinically severe hemophilia A
4. Previous exposure to FVIII therapy
5. No prior history of hypersensitivity or anaphylaxis associated with an FVIII or intravenous immunoglobulin administration.
6. No measurable inhibitor against FVIII
7. Willing to participate and receive treatment in a future Spark hemophilia A gene therapy study.

Exclusion Criteria:

1. Documented active hepatitis B or C within the past 12 months of Screening
2. Currently on antiviral therapy to treat hepatitis B or C;
3. Documented significant liver disease within the past 6 months of Screening
4. Have serological evidence of HIV-1 or HIV-2
5. Anti-AAV-Spark 200 neutralizing titers ≥1:1
6. Previously received SPK-8011;
7. Previously dosed with any investigational or approved gene therapy product at any time or treated with an investigational drug within the last 12 weeks;
8. Planned surgical procedure in the next 12 months requiring FVIII prophylactic treatment.
9. Any history of chronic infection or other chronic disease, concurrent clinically significant major disease (such as liver abnormalities or type I diabetes) including active malignancy, except for non-melanoma skin cancer, any other condition or any other unspecified reasons that, in opinion of the Investigator or Sponsor, makes the participant unsuitable for participation and dosing in a future clinical study for Spark's hemophilia A gene therapy.
10. Unable or unwilling to comply with the schedule of visits and/or study assessments described in the protocol.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetically male
Study Population: Adult males with clinically severe hemophilia A (i.e., ≤2% IU/dL FVIII activity level), who meet eligibility criteria for neutralizing antibody (NAb) to AAV-Spark200.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Number of bleeding events, annualized | 12 months
  Annualized bleeding rate (ABR)

SECONDARY OUTCOMES:
Dose and total FVIIII consumption | 12 months
  Total FVIII replacement therapy consumption and the corresponding dose
Annualized number of infusions (AIR) | 12 months
  Number of reported infusions over the study period

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Bloodworks Northwest, Seattle, Washington
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Austrailia
- Canada (2):
  - Providence Hematology/St. Paul's Hosptial, Vancouver, British Columbia
  - McMaster University / Royal Prince Alfred Hospital, Hamilton, Ontario
- Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No